CLINICAL TRIAL: NCT02660294
Title: Intrauterine Autologous Platelet -Enriched Plasma Infusion Compared to Hormonal Replacement Therapy for Enhancing Endometrial Thickness in Patients Undergoing ICSI
Brief Title: Intrauterine Autologous PRP Infusion Compared to HRT for Enhancing Endometrial Thickness in Patients Undergoing ICSI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, rasha medhat abdul-hady, DR. Rasha Medhat Abdul-hady, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP-IVF
Record Dates: First submitted 2016-01-16; First posted 2016-01-21 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platlet rich plasma (Experimental): For those with endometrial thickness less than 7 mm intrauterine injection of platlet rich plasma (PRP) for enhancing endometrial thickness and receptivity
  Interventions: Biological: platlet rich plasma
- Hormone replacement therapy (No Intervention): Oral intake of estradiol valerate for those with endometrial thickness less than 7 mm will improve endometrial receptivity

INTERVENTIONS:
Biological: platlet rich plasma — Platelet-rich plasma (PRP) is prepared from fresh whole blood which is collected from a peripheral vein, stored in acid citrate dextrose solution A (ACD-A) anticoagulant and processed to increase platelets by separating various components of blood
  Arms: Platlet rich plasma

SUMMARY:
Successful embryo implantation needs an optimum embryonic development with a receptive endometrium. Endometrial thickness is an independant factor for endometrial receiptivity. The aim of that trial is to assess the benefecial effect of platelt rich plasma in copmarison with standard hormonal therapy.

DETAILED DESCRIPTION:
This is a single blinded randomized trial comparing the effect of of platlet rich plasma versus hormonal therapy on endometrial thickness and consequently endometrial receptivity. The primary endpoint of this trial is clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ICSI
* endometrial thickness less than 7 mm on early follicular phase

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness in mm | 72 hours
  using transvaginal ultrasound to measure endometrial thickness in mm

SECONDARY OUTCOMES:
clinical pregnancy rate | 4 weeks after embryo transfer
  using transvaginal ultrasound to detect fetal cardiac activity

CONTACTS AND LOCATIONS:
Overall Officials: RASHA DR MEDHAT, MD, Principal Investigator — Ain Shams University
Locations (1):
- Rasha, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided